CLINICAL TRIAL: NCT01711645
Title: Phase IV, Open Label Trial to Evaluate Immunogenicity of Tdap Vaccine in Post-Partum Women to Optimize Vaccination Schedule for Women Who May Have a Subsequent Child
Brief Title: Tdap Vaccine in Post-Partum Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Prevention
Other Study IDs: 11-0035; HHSN272201300023I
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2015-04-08

CONDITIONS: Diphtheria; Pertussis; Tetanus
Keywords: Acellular; Adacel®; Diptheria toxoids; Pertussis; postpartum; Tdap; Tetanus; women
MeSH Terms: conditions — Diphtheria; Whooping Cough; Tetanus | interventions — Tetanus Toxoid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adacel® Tdap vaccine (Experimental): 55 postpartum subjects receive a single intramuscular (IM) 0.5 mL dose of Adacel® (Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed).
  Interventions: Biological: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed onto aluminum phosphate

INTERVENTIONS:
Biological: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed onto aluminum phosphate — 55 postpartum subjects receive a single intramuscular (IM) 0.5 mL dose of Adacel® (Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed).

SUMMARY:
Monitoring immune response and longevity in serum and milk after Tdap administration to postpartum women. The clinical trial will involve women (aged 18 - 45 years) who have just delivered full-term infants (greater than or equal to 37 completed weeks of gestation) at Vanderbilt University Medical Center. The enrollment period will be fifteen months. The duration is over two years of observation.

DETAILED DESCRIPTION:
This is a single site, prospective study involving only one intervention, receipt of a single 0.5 mL intramuscular (IM) dose of Adacel (Tetanus toxoid, reduced diphtheria toxoid and acellular Pertussis) vaccine, among 55 healthy post partum women. The purpose of the study is to examine the immune responses and subsequent decline in serum and breast milk antibody titers over two years of observation. The clinical trial will involve women (aged 18 - 45 years) who have just delivered full-term infants (greater than or equal to 37 completed weeks of gestation) at Vanderbilt University Medical Center. One particular population at Vanderbilt to target will be the "centering prenatal care group" that has breastfeeding rates as high as 75 percent at hospital discharge and maintained at 20 percent at 6 months. The enrollment period will be fifteen months. The subjects, staff assessing subjects, and laboratory personnel will be aware of receipt of the vaccine. Since only a single vaccine product is being utilized, there is no blinding needed of the subjects or staff.

ELIGIBILITY:
Inclusion Criteria:

-Healthy, postpartum women as determined by medical history aged 18 - 45 years of age inclusive. -Women 1-4 days postpartum from delivery of full-term infants. Full-term will be defined as estimated gestational age of greater than or equal to 37 completed weeks of pregnancy determined by menstrual dating and concordant with ultrasound findings as per ACOG bulletin #101). -Provide written informed consent prior to initiation of any study procedures. -Available for the entire study period. -Able to understand and complete all relevant study procedures during study participation (women who ultimately have limited ability to breast feed after enrollment will not be excluded from the study).

Exclusion Criteria:

-Prior receipt of a tetanus or diphtheria-containing vaccine within two years of enrollment. -Prior receipt of a tetanus and diphtheria toxoid and acellular pertussis vaccine within two years of enrollment. -Known or suspected impairment of immunologic function. -Febrile illness within the last 24 hours or an oral temperature >/= 100.4 degrees F (>/= 38 degrees C) at the time of enrollment. -History of documented tetanus, diphtheria, or pertussis disease within the preceding 5 years. -History of allergic or adverse reaction to diphtheria, tetanus, or pertussis vaccines. -Receipt of any steroids, immunoglobulins, other blood products/transfusion within the past six months- excluding Rh immunoglobulin (Rhogam™ and Rhophylac™). -Is enrolled or plans to enroll in another clinical trial with an investigational product while participating in this study (observational studies are allowed). -Known active infection with HIV, hepatitis B, or hepatitis C. -History of alcohol or drug abuse in the last 5 years. -Any condition which, in the opinion of the investigators, may pose a health risk to the subject or interfere with the evaluation of the study objectives. -Any woman with health condition who is currently taking glucocorticoids, i.e., oral, parenteral, and high-dose inhaled steroids, and immunosuppressive or cytotoxic drugs. -Sensitive to latex, based on package insert -Progressive or unstable neurologic condition, based on package insert. -Receipt of influenza or other vaccines concomitantly administered or for 42 days following Adacel, based on package insert.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2012-10-26 (Actual); Primary Completion 2015-08-28 (Actual); Study Completion 2015-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postpartum participants were recruited within 1-4 days of full-term delivery in the Nashville area between 26Oct2012 and 03Sep2013.
Groups:
- Adacel® Tdap Vaccine: Postpartum participants receive a single intramuscular (IM) 0.5 mL dose of Adacel® (Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed) as a single intramuscular (IM) 0.5 mL dose
Period: Overall Study
Arm/Group | Adacel® Tdap Vaccine
Started | 55
Completed | 36
Not Completed | 19
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 6
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise in Serum Immunoglobulin G (IgG) by ELISA at Week 2
Description: Blood was collected from participants at baseline prior to vaccination and at 2 weeks after vaccination for assessment of IgG by ELISA against the pertussis toxin (PT), filamentous hemaggluttinin (FHA), pertactin (PRN) and fimbrae (FIM) antigens. Antibody concentrations were reported as ELISA units per milliliter (EU/mL). The geometric mean of participants' fold rise in antibody concentrations from baseline to post vaccination was calculated, along with the 95% confidence interval (CI).
Time Frame: Prior to and 2 weeks following vaccination
Population: All participants with specimens collected and data reported for baseline and the post-vaccination timepoint were included in the analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 52
Fold Rise
  PT | 4.8 [3.8 to 5.9]
  FHA | 8.6 [7.2 to 10.4]
  PRN | 21.6 [14.4 to 32.5]
  FIM | 22.4 [12.4 to 40.5]

2. Primary Outcome: Geometric Mean Fold Rise in Serum IgG by ELISA at Week 6
Description: Blood was collected from participants at baseline prior to vaccination and at 6 weeks after vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. The geometric mean of participants' fold rise in antibody concentrations from baseline to post vaccination was calculated, along with the 95% CI.
Time Frame: Prior to and 6 weeks following vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 53
Fold Rise
  PT | 3.5 [2.9 to 4.4]
  FHA | 6.7 [5.7 to 8.0]
  PRN | 19.1 [12.5 to 29.1]
  FIM | 18.6 [11.1 to 31.1]

3. Primary Outcome: Geometric Mean Fold Rise in Serum IgG by ELISA at Month 6
Description: Blood was collected from participants at baseline prior to vaccination and at 6 months after vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. The geometric mean of participants' fold rise in antibody concentrations from baseline to post vaccination was calculated, along with the 95% CI.
Time Frame: Prior to and 6 months following vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 49
Fold Rise
  PT | 1.9 [1.6 to 2.3]
  FHA | 3.4 [3.0 to 3.9]
  PRN | 8.1 [5.5 to 12.0]
  FIM | 10.1 [6.2 to 16.3]

4. Primary Outcome: Geometric Mean Fold Rise in Serum IgG by ELISA at Month 12
Description: Blood was collected from participants at baseline prior to vaccination and at 12 months after vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. The geometric mean of participants' fold rise in antibody concentrations from baseline to post vaccination was calculated, along with the 95% CI.
Time Frame: Prior to and 12 months following vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 48
Fold Rise
  PT | 1.6 [1.4 to 1.9]
  FHA | 2.5 [2.2 to 2.8]
  PRN | 5.1 [3.6 to 7.1]
  FIM | 6.9 [4.3 to 11.0]

5. Primary Outcome: Geometric Mean Fold Rise in Serum IgG by ELISA at Month 18
Description: Blood was collected from participants at baseline prior to vaccination and at 18 months after vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. The geometric mean of participants' fold rise in antibody concentrations from baseline to post vaccination was calculated, along with the 95% CI.
Time Frame: Prior to and 18 months following vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 46
Fold Rise
  PT | 1.6 [1.4 to 1.8]
  FHA | 2.4 [2.1 to 2.8]
  PRN | 4.6 [3.3 to 6.4]
  FIM | 6.8 [4.3 to 10.8]

6. Primary Outcome: Geometric Mean Fold Rise in Serum IgG by ELISA at Month 24
Description: Blood was collected from participants at baseline prior to vaccination and at 24 months after vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. The geometric mean of participants' fold rise in antibody concentrations from baseline to post vaccination was calculated, along with the 95% CI.
Time Frame: Prior to and 24 months following vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 35
Fold Rise
  PT | 1.4 [1.2 to 1.6]
  FHA | 2.2 [1.9 to 2.5]
  PRN | 4.9 [3.3 to 7.4]
  FIM | 7.0 [4.0 to 12.2]

7. Primary Outcome: ELISA Geometric Mean Concentrations (GMC) of Serum IgG to PT, FHA, PRN and FIM at Baseline
Description: Blood was collected from participants at baseline prior to vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. Antibody concentrations were reported as ELISA units per milliliter (EU/mL). A value of 5 EU/mL was imputed for results reported as below the lower limit of quantitation (LLOQ) (<10 EU/mL). The geometric mean of participants' concentrations at the timepoint was calculated, along with the 95% CI.
Time Frame: Baseline (prior to vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 55
EU/mL
  PT | 6.6 [5.7 to 7.7]
  FHA | 15.9 [12.6 to 20.1]
  PRN | 20.3 [14.1 to 29.2]
  FIM | 38.1 [23.4 to 62.1]

8. Primary Outcome: ELISA GMCs of Serum IgG to PT, FHA, PRN and FIM at Week 2
Description: Blood was collected from participants at 2 weeks after vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. A value of 5 EU/mL was imputed for results reported as below LLOQ. The geometric mean of participants' concentrations at the timepoint was calculated, along with the 95% CI.
Time Frame: 2 weeks post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 52
EU/mL
  PT | 51.5 [39.2 to 67.7]
  FHA | 154.3 [132.3 to 179.9]
  PRN | 581.5 [430.4 to 785.6]
  FIM | 1156.3 [794.2 to 1683.5]

9. Primary Outcome: ELISA GMCs of Serum IgG to PT, FHA, PRN and FIM at Week 6
Description: Blood was collected from participants at 6 weeks after vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. A value of 5 EU/mL was imputed for results reported as below LLOQ. The geometric mean of participants' concentrations at the timepoint was calculated, along with the 95% CI.
Time Frame: 6 weeks post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 53
EU/mL
  PT | 37.5 [28.5 to 49.3]
  FHA | 126.1 [106.5 to 149.2]
  PRN | 496.8 [355.6 to 694.1]
  FIM | 905.1 [663.2 to 1235.2]

10. Primary Outcome: ELISA GMCs of Serum IgG to PT, FHA, PRN and FIM at Month 6
Description: Blood was collected from participants at 6 months after vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. A value of 5 EU/mL was imputed for results reported as below LLOQ. The geometric mean of participants' concentrations at the timepoint was calculated, along with the 95% CI.
Time Frame: 6 months post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 49
EU/mL
  PT | 19.2 [15.0 to 24.6]
  FHA | 62.4 [53.3 to 73.0]
  PRN | 212.3 [149.9 to 300.9]
  FIM | 492.8 [358.4 to 677.6]

11. Primary Outcome: ELISA GMCs of Serum IgG to PT, FHA, PRN and FIM at Month 12
Description: Blood was collected from participants at 12 months after vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. A value of 5 EU/mL was imputed for results reported as below LLOQ. The geometric mean of participants' concentrations at the timepoint was calculated, along with the 95% CI.
Time Frame: 12 months post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 48
EU/mL
  PT | 15.1 [11.6 to 19.6]
  FHA | 46.2 [39.0 to 54.8]
  PRN | 141.1 [103.4 to 192.6]
  FIM | 368.7 [264.2 to 514.5]

12. Primary Outcome: ELISA GMCs of Serum IgG to PT, FHA, PRN and FIM at Month 18
Description: Blood was collected from participants at 18 months after vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. A value of 5 EU/mL was imputed for results reported as below LLOQ. The geometric mean of participants' concentrations at the timepoint was calculated, along with the 95% CI.
Time Frame: 18 months post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 46
EU/mL
  PT | 15.1 [12.0 to 19.1]
  FHA | 44.6 [35.4 to 56.2]
  PRN | 121.1 [84.0 to 174.5]
  FIM | 330.7 [234.6 to 466.1]

13. Primary Outcome: ELISA GMCs of Serum IgG to PT, FHA, PRN and FIM at Month 24
Description: Blood was collected from participants at 24 months after vaccination for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens. A value of 5 EU/mL was imputed for results reported as below LLOQ. The geometric mean of participants' concentrations at the timepoint was calculated, along with the 95% CI.
Time Frame: 24 months post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 35
EU/mL
  PT | 10.8 [7.9 to 14.6]
  FHA | 39.0 [30.1 to 50.6]
  PRN | 114.1 [74.9 to 173.9]
  FIM | 298.0 [187.3 to 474.0]

14. Primary Outcome: Count of Participants With 4-fold Rise in ELISA Antibody Concentrations at Week 2
Description: Blood samples were collected from participants for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens at baseline prior to vaccination and 2 weeks after vaccination. A 4-fold rise in antibody concentration from prior to vaccination was defined as a post-vaccination IgG greater than or equal to 40 EU/mL for participants with baseline IgG concentrations less than the LLOQ (10), or 4 times the baseline IgG concentration for baseline IgG concentrations greater than the LLOQ.
Time Frame: Prior to and 2 weeks after vaccination
Population: All participants with blood collected and results reported at both timepoints are included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 52
Participants
  PT | 31
  FHA | 45
  PRN | 43
  FIM | 34

15. Primary Outcome: Count of Participants With 4-fold Rise in ELISA Antibody Concentrations at Week 6
Description: Blood samples were collected from participants for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens at baseline prior to vaccination and 6 weeks after vaccination. A 4-fold rise in antibody concentration from prior to vaccination was defined as a post-vaccination IgG greater than or equal to 40 EU/mL for participants with baseline IgG concentrations less than the LLOQ (10), or 4 times the baseline IgG concentration for baseline IgG concentrations greater than the LLOQ.
Time Frame: Prior to and 6 weeks after vaccination
Population: All participants with blood collected and results reported at both timepoints are included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 53
Participants
  PT | 21
  FHA | 44
  PRN | 42
  FIM | 34

16. Primary Outcome: Count of Participants With 4-fold Rise in ELISA Antibody Concentrations at Month 6
Description: Blood samples were collected from participants for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens at baseline prior to vaccination and 6 months after vaccination. A 4-fold rise in antibody concentration from prior to vaccination was defined as a post-vaccination IgG greater than or equal to 40 EU/mL for participants with baseline IgG concentrations less than the LLOQ (10), or 4 times the baseline IgG concentration for baseline IgG concentrations greater than the LLOQ.
Time Frame: Prior to and 6 months after vaccination
Population: All participants with blood collected and results reported at both timepoints are included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 49
Participants
  PT | 5
  FHA | 18
  PRN | 34
  FIM | 29

17. Primary Outcome: Count of Participants With 4-fold Rise in ELISA Antibody Concentrations at Month 12
Description: Blood samples were collected from participants for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens at baseline prior to vaccination and 12 months after vaccination. A 4-fold rise in antibody concentration from prior to vaccination was defined as a post-vaccination IgG greater than or equal to 40 EU/mL for participants with baseline IgG concentrations less than the LLOQ (10), or 4 times the baseline IgG concentration for baseline IgG concentrations greater than the LLOQ.
Time Frame: Prior to and 12 months after vaccination
Population: All participants with blood collected and results reported at both timepoints are included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 48
Participants
  PT | 5
  FHA | 5
  PRN | 28
  FIM | 26

18. Primary Outcome: Count of Participants With 4-fold Rise in ELISA Antibody Concentrations at Month 18
Description: Blood samples were collected from participants for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens at baseline prior to vaccination and 18 months after vaccination. A 4-fold rise in antibody concentration from prior to vaccination was defined as a post-vaccination IgG greater than or equal to 40 EU/mL for participants with baseline IgG concentrations less than the LLOQ (10), or 4 times the baseline IgG concentration for baseline IgG concentrations greater than the LLOQ.
Time Frame: Prior to and 18 months after vaccination
Population: All participants with blood collected and results reported at both timepoints are included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 46
Participants
  PT | 3
  FHA | 7
  PRN | 25
  FIM | 26

19. Primary Outcome: Count of Participants With 4-fold Rise in ELISA Antibody Concentrations at Month 24
Description: Blood samples were collected from participants for assessment of IgG by ELISA against the PT, FHA, PRN and FIM antigens at baseline prior to vaccination and 24 months after vaccination. A 4-fold rise in antibody concentration from prior to vaccination was defined as a post-vaccination IgG greater than or equal to 40 EU/mL for participants with baseline IgG concentrations less than the LLOQ (10), or 4 times the baseline IgG concentration for baseline IgG concentrations greater than the LLOQ.
Time Frame: Prior to and 24 months after vaccination
Population: All participants with blood collected and results reported at both timepoints are included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 35
Participants
  PT | 1
  FHA | 2
  PRN | 19
  FIM | 20

20. Primary Outcome: Kinetics of the ELISA IgG Antibody Rise in Serum
Description: The assessment of the kinetics of the ELISA IgG antibody rise in serum was defined by the protocol as the geometric mean fold rise at each timepoint (reported separately above). No additional analysis was pre-defined or performed for this outcome measure.
Time Frame: Prior to and following Tdap, through 24 months post-vaccination
Population: No analysis was conducted for this outcome measure. See previous outcome measures for geometric mean fold rises at each timepoint.
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 0

21. Secondary Outcome: ELISA GMC of Breast Milk IgA to Pertussis Toxin (PT) at Baseline.
Description: Breast milk (colostrum) was collected from participants at baseline prior to vaccination for assessment of secretory IgA (sIgA) to the PT antigen by ELISA. Available data at the timepoint were summarized by geometric mean of the concentration as reported in EU/mL along with the 95% confidence interval. The lower limit of quantitation (LLOQ) of the assay was 10. Results of <10 were reported as half the LLOQ (5).
Time Frame: Baseline (prior to vaccination)
Population: All participants providing a breast milk (colostrum) sample at the timepoint are included in the analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 4
EU/mL | 28.8 [2.5 to 336.9]

22. Secondary Outcome: ELISA GMC of Breast Milk IgA to PT at Week 2
Description: Breast milk was collected from participants at 2 weeks after vaccination for assessment of secretory IgA (sIgA) to PT and FHA by ELISA. Available data at the timepoint were summarized by geometric mean of the concentration as reported in EU/mL. Note that for the PT at this timepoint, all participants had a value of 5, the imputed value for below the LLOQ of the assay (<10), and so the 95% CI is not reported, as there was no measurable variability in the data. The range is reported.
Time Frame: 2 weeks post vaccination
Population: All participants providing a breast milk sample at the timepoint are included in the analysis population.
Measure: Geometric Mean (Full Range); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 34
EU/mL | 5.0 [5.0 to 5.0]

23. Secondary Outcome: ELISA GMC of Breast Milk IgA to PT at Week 6
Description: Breast milk was collected from participants at 6 weeks after vaccination for assessment of secretory IgA (sIgA) to PT and FHA by ELISA. Available data at the timepoint were summarized by geometric mean of the concentration as reported in EU/mL. Note that for the PT at this timepoint, all participants had a value of 5, the imputed value for below the LLOQ of the assay (<10), and so the 95% CI is not reported, as there was no measurable variability in the data. The range is reported.
Time Frame: 6 weeks post vaccination
Population: All participants providing a breast milk sample at the timepoint are included in the analysis population.
Measure: Geometric Mean (Full Range); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 35
EU/mL | 5.0 [5.0 to 5.0]

24. Secondary Outcome: ELISA GMC of Breast Milk IgA to PT at Month 6
Description: as for outcome 23
Time Frame: 6 months post vaccination
Population: All participants providing a breast milk sample at the timepoint are included in the analysis population.
Measure: Geometric Mean (Full Range); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 22
EU/mL | 5.0 [5.0 to 5.0]

25. Secondary Outcome: ELISA GMC of Breast Milk IgA to FHA at Baseline.
Description: Breast milk (colostrum) was collected from participants at baseline prior to vaccination for assessment of secretory IgA (sIgA) to the FHA antigen by ELISA. Available data at the timepoint were summarized by geometric mean of the concentration as reported in EU/mL along with the 95% confidence interval.
Time Frame: Baseline (prior to vaccination)
Population: All participants providing a breast milk (colostrum) sample at the timepoint are included in the analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 4
EU/mL | 28.3 [6.9 to 116.6]

26. Secondary Outcome: ELISA GMC of Breast Milk IgA to FHA at Week 2.
Description: Breast milk was collected from participants at 2 weeks post vaccination for assessment of secretory IgA (sIgA) to the FHA antigen by ELISA. Available data at the timepoint were summarized by geometric mean of the concentration as reported in EU/mL along with the 95% confidence interval.
Time Frame: 2 weeks post vaccination
Population: All participants providing a breast milk sample at the timepoint are included in the analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 34
EU/mL | 5.4 [4.8 to 6.0]

27. Secondary Outcome: ELISA GMC of Breast Milk IgA to FHA at Week 6.
Description: Breast milk was collected from participants at 6 weeks post vaccination for assessment of secretory IgA (sIgA) to the FHA antigen by ELISA. Available data at the timepoint were summarized by geometric mean of the concentration as reported in EU/mL. Note that for the FHA at this timepoint, all participants had a concentration of 5, the imputed value for below the LLOQ of the assay (<10), and so the 95% CI is not reported, as there was no measurable variability in the data. The range is reported.
Time Frame: 6 weeks post vaccination
Population: All participants providing a breast milk sample at the timepoint are included in the analysis population.
Measure: Geometric Mean (Full Range); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 35
EU/mL | 5.0 [5.0 to 5.0]

28. Secondary Outcome: ELISA GMC of Breast Milk IgA to FHA at Month 6.
Description: Breast milk was collected from participants at 6 months post vaccination for assessment of secretory IgA (sIgA) to the FHA antigen by ELISA. Available data at the timepoint were summarized by geometric mean of the concentration as reported in EU/mL along with the 95% confidence interval.
Time Frame: 6 months post vaccination
Population: All participants providing a breast milk sample at the timepoint are included in the analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 22
EU/mL | 5.2 [4.8 to 5.8]

29. Secondary Outcome: ELISA GMC of Breast Milk IgA to PRN and FIM by Study Day.
Description: Breast milk (colostrum) was collected from participants at baseline prior to vaccination for assessment of secretory IgA (sIgA) to the PRN and FIM antigen by ELISA. Available data at the timepoint were to be summarized by geometric mean of the concentration as reported in EU/mL along with the 95% confidence interval. The lower limit of quantitation (LLOQ) of the assay was 10 EU/mL.
Time Frame: Baseline (prior to vaccination), Week 2, Week 6 and Month 6 post vaccination
Population: The laboratory staff was not successful in attempts to conduct the ELISA assay against the pertactin and fimbrae antigens with the breast milk samples.
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 0

30. Secondary Outcome: Proportion of Participants With 4-fold Rise in Antibody in Breast Milk by Study Day.
Description: Breast milk samples were collected from participants for evaluation of PT and FHA secretory IgA (sIgA) by ELISA. The lower limit of quantification (LLOQ) for the assay was 10 EU/mL. A 4-fold rise in concentration from prior to vaccination was defined as a post-vaccination sIgA concentration greater than or equal to 40 EU/mL for participants with baseline sIgA concentrations less than the LLOQ, or 4 times the baseline sIgA concentration for baseline sIgA concentrations greater than the LLOQ.
Time Frame: Prior to vaccination, 2 weeks, 6 weeks, and 6 months after vaccination
Population: Only 4 participants were able to provide a breast milk (colostrum) sample at baseline and post vaccination samples had no detectable titer, resulting in a fold-rise analysis being uninterpretable; therefore, this analysis was not conducted.
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 0

31. Secondary Outcome: Geometric Mean Fold Rise in Antibody Concentrations Assessed by ELISA in Breast Milk by Study Day
Description: Breast milk samples were collected from participants for evaluation of secretory IgA (sIgA) by ELISA. Geometric mean fold rise was defined as the geometric mean of participants' fold rise in post vaccination sIgA relative to the pre-vaccination sIgA.
Time Frame: Prior to vaccination, 2 weeks, 6 weeks, and 6 months after vaccination
Population: as for outcome 30
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 0

32. Secondary Outcome: Kinetics of the ELISA IgG Antibody Decline in Breast Milk Expressed in EU/ml.
Description: Breast milk samples were collected from participants for evaluation of PT and FHA secretory IgA (sIgA) by ELISA. The protocol defined kinetics as assessment at each post-vaccination timepoint of the geometric mean fold rise, defined as the geometric mean of participants' fold rise in post vaccination sIgA relative to the pre-vaccination sIgA.
Time Frame: Prior to vaccination, 2 weeks, 6 weeks, and 6 months after vaccination
Population: as for outcome 30
Arm/Group | Adacel® Tdap Vaccine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Since pertussis vaccine is offered as standard of care to healthy adults, including postpartum women, anticipated AEs related to pertussis vaccine administration, as per Package Insert, were not collected. AEs reported for this protocol were limited to 1. severe vaso-vagal reaction, including loss of consciousness or > grade 2 hypotension, associated with the blood draw; and 2. adverse events leading to infection or inability to breast feed following the use of the breast pump.
Description: Anticipated adverse events related to administration of the pertussis vaccine as per Package Insert include injection site reactions (pain, swelling and erythema) and systemic reactions (headache body ache and muscle weakness). Events meeting VAERS reporting requirements were to be reported to VAERS and not collected for this protocol.
Arm/Group | Adacel® Tdap Vaccine
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less